CLINICAL TRIAL: NCT03860662
Title: Doctor, Physical Medicine and Rehabilitation
Brief Title: The Effect of Oral Baclofen and Botulinum Toxin Treatments in Hemiplegic Spasticity on the Nociceptive Flexor Reflex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, ERTURK GUNTURK, research assistant doctor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MustafaKUPMR
Record Dates: First submitted 2019-02-08; First posted 2019-03-04 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Stroke Sequelae; Spastic Hemiplegia
Keywords: Antispastic drugs; Nociceptive flexor reflex; Baclofen; Botulinum toxin
MeSH Terms: conditions — Hemiplegia | interventions — Botulinum Toxins, Type A; Baclofen

STUDY DESIGN:
Intervention Model Description: The purpose of this thesis is to research the effect of oral baclofen treatment and botulinum toxin injection treatments over the electromyographic nociceptive flexor reflex (NFR) threshold in hemiplegic patients with spasticity. The results of the study evaluated the Modified Ashworth Scale, joint range of motion, muscle strength, Brunnstrom stages, Barthel daily life activities index, electromyographic nociceptive flexor reflex (NFR) threshold.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Spastic hemiplegia , Botox (Active Comparator): Botulinum toxin (BTX), being one of the most potent biological toxins, acts by blocking neuromuscular transmission via inhibiting acetylcholine release. Currently, focal spasticity is being treated successfully with BTX via injecting in the spastic muscles( Dose: 300-400 iu). Two antigenically distinct serotypes of BTX are available on the market as type A and B.
  Interventions: Diagnostic Test: Nociceptor flexor reflex; Drug: Botox
- Spastic hemiplegia, Baclofen (Other): Baclofen is an agonist that has presynaptic and postsynaptic effects on monosynaptic and polysynaptic pathways by binding to GABA B receptors. The recommended dosing regimen is initiated with 5 mg 3 times a day. It can be increased by 15-mg/d increments at 3-day intervals as needed. Dosing should not exceed 80 mg/d.
  Interventions: Diagnostic Test: Nociceptor flexor reflex; Drug: Baclofen

INTERVENTIONS:
Diagnostic Test: Nociceptor flexor reflex — The nociceptive flexion reflex (NFR) is a physiological, polysynaptic reflex allowing for painful stimuli to activate an appropriate withdrawal response
Drug: Botox — botox
  Arms: Spastic hemiplegia , Botox
Drug: Baclofen — baclofen
  Arms: Spastic hemiplegia, Baclofen

SUMMARY:
The purpose of this thesis is to research the effect of oral baclofen treatment and botulinum toxin injection treatments over the electromyographic nociceptive flexor reflex (NFR) threshold in hemiplegic patients with spasticity. The results of the study evaluated the Modified Ashworth Scale, joint range of motion, muscle strength, Brunnstrom stages, Barthel daily life activities index, electromyographic nociceptive flexor reflex (NFR) threshold.

DETAILED DESCRIPTION:
Spasticity is defined as increased resistance tied to speed against passive movements and is related to hyperactive reflexes after upper motor neuron lesions. The hemiplegia table, which develops after subsiding, brings many problems along with it. Spasticity is one of these problems. Spasticity frequently leads to difficulty in the activities of daily life. It delays functional recovery, causes pain, and leads to secondary complications.

The objective of spasticity treatment minimizes the negative effects of hypertension without endangering function. Systematic medication treatment (baclofen, diazepam, dantrolen, and tizanidine) or local treatment (botulinum toxin, phenyl injection) are administered in spasticity treatment. The botulinum toxin prevents the secretion of acetylcholine in nerve endings and creates a presynaptic neuromuscular block. There are numerous studies that show that botulinum toxin is effective in spasticity.

Baclofen is a gamma aminobutyric acid (GABA) agonist. It passes through the blood-brain barrier and binds to the GABAb receptors of the spinal cord. Baclofen decreases spasms, clonus, and resistance to germs.

Various studies of electrophysiological reflexes are conducted to evaluate spasticity and to study neuronal circuits. The electrophysiological test is a tool used in studying the changes in spinal cord function and spinal reflexes in patients. The flexor reflex known as the recoil reflex is a polysynaptic and multisegmental reflex. It provides for avoidance and protection from internal and external stimulants that may be harmful for the body.

The purpose of the study is to research the effect of oral baclofen treatment and botulinum toxin injection treatments over the electromyographic nociceptive flexor reflex (NFR) threshold in hemiplegic patients with spasticity.

PURPOSE OF THE RESEARCH The purpose of this thesis is to research the effect of oral baclofen treatment and botulinum toxin injection treatments over the electromyographic nociceptive flexor reflex (NFR) threshold in hemiplegic patients with spasticity. The results of the study evaluated the Modified Ashworth Scale, joint range of motion, muscle strength, Brunnstrom stages, Barthel daily life activities index, electromyographic nociceptive flexor reflex (NFR) threshold

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-60
* To accept voluntary participation in the study
* Spastic Hemiplegia (Modified Ashworth Scale 2 and above)

Exclusion Criteria:

* Pregnant women, breastfeeding and younger than 18 years
* To have medication and substance use causing neuropathy in the history of the disease and / or neuropathy
* Companies that have received botulinum toxin injection therapy and / or oral antispastic therapy within the last 6 months
* Have a history of allergies and hypersensitivity to usability drug
* Injection treatment planned purification hematoma, cleaning or skin lesion to be

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2018-05-26 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-04-21 (Actual)

PRIMARY OUTCOMES:
thershold of nociceptive flexor reflex | 6 weeks
  The nociceptive flexion reflex (NFR) is a physiological, polysynaptic reflex allowing for painful stimuli to activate an appropriate withdrawal response
Barthel index | 6 weeks
  The Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e. feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. The index also indicates the need for assistance in care.The final score on the Barthel index ranges from 0, or complete dependence, to 100, or complete independence .
Vısual analog scale | 6 weeks
  When using a VAS to assess pain, subjects are asked to indicate intensity by marking a (usually) 100-mm-long horizontal line that is labeled "no pain" at one end and "worst pain possible" at the other end. This requires the patient to be able to equate the length of the line (as measured from the left-hand side to the point marked) with the amount of pain they are experiencing. Higher values represent worse outcome.
Range of motion | 6 weeks
  Range of motion (ROM) is the measurement of the amount of movement around a specific joint or body part
Modified Ashworth scale | 6 weeks
  The Modified Ashworth scale (MAS) measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. Higher values represent worse outcome.
  (0) No increase in muscle tone
  (1) Slight increase in muscle tone, manifested by a catch and release or byminimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension.(1+) Slight increase in muscle tone, manifested by a catch, followed by minimalresistance throughout the remainder (less than half) of the ROM.(2) More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved.(3) Considerable increase in muscle tone, passive movement difficult.(4) Affected part(s) rigid in flexion or extension

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided